CLINICAL TRIAL: NCT00534027
Title: A Phase 1b/2 Study of AMG 655 in Combination With Paclitaxel and Carboplatin for the First-Line Treatment of Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060295
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Non-Small Cell Lung Cancer; Paclitaxel; Carboplatin; AMG 655
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — conatumumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Arm 2 (Experimental): Low Dose AMG 655 with paclitaxel/carboplatin
  Interventions: Drug: AMG 655
- Arm 3 (Placebo Comparator): Placebo with paclitaxel/carboplatin
  Interventions: Other: AMG 655 placebo
- Arm 1 (Experimental): AMG 655 High doseplus paclitaxel/carboplatin
  Interventions: Drug: AMG 655

INTERVENTIONS:
Drug: AMG 655 — AMG 655 is a monoclonal antibody directed against TR-2.
  Other Names: Placebo
  Arms: Arm 1; Arm 2
Other: AMG 655 placebo — Inactive dummy AMG 655 (to maintain blind)
  Arms: Arm 3

SUMMARY:
Part 1 is complete. Part 2 is a multi-center, randomized, double-blind, placebo-controlled, phase 2 segment that will commence upon identification of the maximum tolerated dose in part 1. The Primary objective of Part 2 of the study is to estimate efficacy in combination with carboplatin and paclitaxel. Subjects will be randomized at a 1:1:1 ratio to 1 of 3 treatment arms. Subjects in each of the 3 arms will receive up to 6 cycles of paclitaxel/carboplatin (at the same dose and schedule in part 1) in combination with either AMG 655 at the maximum tolerated dose (Arm 1), AMG 655 at a lower dose (Arm 2), or AMG 655 placebo (Arm 3) IV Q3W. Randomization will be stratified by ECOG (0 or 1) and disease stage (IIIb or IV/recurrent).

ELIGIBILITY:
Inclusion Criteria:

* Disease Related

  * Histologically or cytologically confirmed non-small cell lung cancer.
  * Subjects must have advanced non-small cell lung cancer defined as stage IIIB with malignant pleural effusion or stage IV or recurrent disease.
  * Planning to receive up to 6 cycles of chemotherapy
  * Eastern Cooperative Oncology Group (ECOG) score of 0 or 1 Demographic
  * Men or women > 18 years of age Ethical
  * Adequate Hematological, renal, hepatic and coagulation function General
  * Plan to begin protocol specific therapy < 7 days after enrollment/randomization

Exclusion Criteria:

* Disease Related

  * Untreated or symptomatic central nervous system metastases. Subjects with a history of brain metastases are eligible if definitive therapy has been administered (surgery and/or radiation therapy), there is no planned treatment for brain metastasis and the subject is clinically stable and off corticosteroids for at least 14 days before enrollment/randomization.
  * Prior chemotherapy as follows:
  * Any prior chemotherapy for advanced non-small cell lung cancer
  * Any prior adjuvant chemotherapy for non-small cell lung cancer < 52 weeks prior to enrollment/randomization. Adjuvant chemotherapy completed > 52 weeks prior to randomization is permitted.
  * Any prior chemoradiation.
  * Central (chest) radiation therapy < 28 days prior to randomization, radiation therapy for peripheral lesions < 14 days prior to enrollment/randomization
  * Other abnormal medical conditions
  * Documented myocardial infarction or unstable/uncontrolled cardiac condition
  * History of arterial thrombosis, pulmonary embolus, deep vein thrombosis or hemorrhagic disorders
  * Major surgical procedure < 30 days prior to enrollment/randomization or not yet recovered from prior major surgery, Minor surgical procedure < 7 days prior to enrollment/randomization or not yet recovered from prior minor surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Until disease progression

SECONDARY OUTCOMES:
Objective response rate, duration of response, time to response, overall survival and incidence of adverse events and clinical laboratory abnormalities | Until disease progression

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Paz-Ares L, Balint B, de Boer RH, van Meerbeeck JP, Wierzbicki R, De Souza P, Galimi F, Haddad V, Sabin T, Hei YJ, Pan Y, Cottrell S, Hsu CP, RamLau R. A randomized phase 2 study of paclitaxel and carboplatin with or without conatumumab for first-line treatment of advanced non-small-cell lung cancer. J Thorac Oncol. 2013 Mar;8(3):329-37. doi: 10.1097/JTO.0b013e31827ce554. PMID 23370314
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com